CLINICAL TRIAL: NCT07341711
Title: Long-term Adaptations of Skeletal Muscle in Overweight and Obese Individuals After Hybrid Training.
Brief Title: Long-term Adaptations of Skeletal Muscle After Hybrid Training.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Ioannis G. Fatouros, Professor, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2482/4.12.2024
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Obesity & Overweight
Keywords: obesity; overweight; high-intensity interval training; skeletal muscle
MeSH Terms: conditions — Obesity; Overweight | interventions — Exercise; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this arm will participate in three hybrid-type HIIT sessions per week over a 6-month period while receiving a balanced diet
  Interventions: Other: Exercise training
- Control group (Active Comparator): Participants in this arm will receive a balanced diet over the 6-month period but will not participate in exercise training
  Interventions: Other: Control group

INTERVENTIONS:
Other: Exercise training — Participants will perform a six-month hybrid training program while receiving a balanced diet. The periodization of hybrid training intervention will consist of three 2-month phases of gradually increased exercise intensity and volume. In every training will participate 5-8 individuals. The training will contain 6-12 different exercises (stations), depending on the phase of the intervention, which will be executed in a circuit for a total of 2-3 rounds, with 2-3 minutes of rest period between sets (depending on the phase). The exercise execution will last 20-45 seconds, and the rest between them will last 30-60 seconds (depending on the phase), while the exercise intensity will range from 75 to 85% of maximal heart rate. The stations of hybrid training will contain multi-joint exercises or neuromuscular activation exercises using either body weight resistance or portable equipment.
  Arms: Intervention group
Other: Control group — Participants will receive a balanced diet but will not participate in any type of exercise training over a six month period.
  Arms: Control group

SUMMARY:
Obesity is a major challenge for public health and renders it imperative to reduce its prevalence. High intensity interval training (HIIT) is a form of exercise training that can efficiently induce weight loss in adults with overweight or obesity, even in the absence of dietary intake manipulation. Hybrid type training represents a form of HIIT, that incorporates both cardiorespiratory and musculoskeletal stimuli, by combining multiple types of exercise into a circuit-type, interval style workout. Recent evidence suggests that long-term participation in hybrid HIIT results in significant health-related benefits. However, the molecular mechanisms driving the chronic effects of hybrid HIIT on cardiometabolic and musculoskeletal health remains to be elucidated.

DETAILED DESCRIPTION:
A total number of 30 adults (both males and females) aged 30-50, meeting the inclusion criteria, will be enrolled in this study. Participants will be randomly assigned to either (i) a Control group or (ii) an Intervention group. The Intervention group will participate in three hybrid-type HIIT sessions per week over a 6-month period while receiving a balanced diet. The Control group will receive a balanced diet over the 6-month period but will not participate in exercise training. At baseline and 6 months, both groups will undergo assessment of their anthropometric profile, body composition, resting metabolic rate, muscle strength and cardiorespiratory capacity and provide resting blood and skeletal muscle samples.

ELIGIBILITY:
Inclusion Criteria:

* BMI: >25 kg/m2 and <40 kg/m2
* Untrained individuals (abstain >1 year from exercise training)
* No dietary intervention over the last 6 months preceding the study
* Low cardiorespiratory fitness level (VO2max: <45 ml/kg/min)
* No use of any medication, dietary supplements
* Low risk for cardiovascular disease
* A weight loss <10% over the last 6 months preceding the study
* Fee of non-communicable diseases (excluding metabolic syndrome)

Exclusion Criteria:

* Low participation rate (<80% completion of the exercise training sessions)
* Unbalanced diet
* Participation in additional exercise training regimes
* Cosumption of anti-inflammatory of pain relief medication

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-08 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Change in mitochondrial size | At baseline and at 6 months
  Mitochondrial size will be measured using transmission electron microscope
Change in mitochondrial density | At baseline and at 6 months
  Mitochondrial density will be measured using transmission electron microscope
Change in mitochondrial count | At baseline and at 6 months
  Mitochondrial count will be determined using transmission electron microscope
Change in mitochondrial distribution | At baseline and at 6 months
  Mitochondrial distribution will be determined using transmission electron microscope
Change in maximum oxygen consumption (VO2max) | At baseline and at 6 months
  Maximum oxygen consumption (VO2max) will be assessed during a cardiopulmonary exercise testing by using a portable indirect calorimetry system
Change in muscle fiber cross-sectional area | At baseline and at 6 months
  Muscle fiber cross-sectional area (μm2) will be measured using immunohistochemical staining for myosin heavy chain
Change in PAX7+ satellite cells count | At baseline and at 6 months
  PAX7+ satellite cells will be determined using immunohistochemistry techniques.
Change in total protein content | At baseline and at 6 months
  Total protein content (total RNA) will be determined in skeletal muscle tissue using real time quantitative-Polymerase Chain Reaction (q-PCR) technique
Change in myonuclei content | At baseline and at 6 months
  Myonuclei content will be determined in skeletal muscle tissue using immunohistochemistry techniques
Change in peroxisome proliferator-activated receptor-gamma coactivator -1a (PGC-1a) expression | At baseline and at 6 months
  PGC-1a expression in skeletal muscle tissue will be assessed using immunoblotting techniques.
Change in Krebs cycle (TCA cycle) enzymes activity | At baseline and at 6 months
  Krebs cycle enzymes activity will be determined using the Seahorse XF Analyzer
Change in protein expression of respiratory chain complexes | At baseline and at 6 months
  Protein expression of respiratory chain complexes will be determined using immunoblotting techniques
Change in cytochrome C oxidase amount and expression | At baseline and at 6 months
  Cytochrome C oxidase amount and expression will be assessed using immunohistochemistry and immunoblotting techniques
Change in ATP synthase amount and expression | At baseline and at 6 months
  ATP synthase amount and expression will be assessed using immunohistochemistry and immunoblotting techniques
Change in citrate synthase amount and expression | At baseline and at 6 months
  Citrate synthase amount and expression will be assessed using immunohistochemistry and immunoblotting techniques
Change in succinate dehydrogenase amount and expression | At baseline and at 6 months
  Succinate dehydrogenase amount and expression will be assessed using immunohistochemistry and immunoblotting techniques
Change in NADH dehydrogenase amount and expression | At baseline and at 6 months
  NADH dehydrogenase amount and expression will be assessed using immunohistochemistry and immunoblotting techniques
Change in mitochondrial oxygen consumption rate | At baseline and at 6 months
  Mitochondrial oxygen consumption rate will be determined using the Seahorse XF Analyzer
Change in spare respiratory capacity | At baseline and at 6 months
  Spare respiratory capacity will be determined using the Seahorse XF Analyzer
Change in mitochondrial maximal respiration | At baseline and at 6 months
  Maximal mitochondrial respiration will be determined using the Seahorse XF Analyzer
Change in mitochondrial basal respiration | At baseline and at 6 months
  Mitochondrial basal respiration will be determined using the Seahorse XF Analyzer
Change in non-mitochondrial respiration | At baseline and at 6 months
  Non-mitochondrial respiration will be determined using the Seahorse XF Analyzer
Change in body fat percentage | At baseline and at 6 months
  Body fat percentage will be assessed using dual energy x-ray absorptiometry (DEXA)
Change in diastolic arterial pressure | At baseline and at 6 months
  Diastolic blood pressure will be measured using a sphygmomanometer

SECONDARY OUTCOMES:
Change in density and distribution of capillaries | At baseline and at 6 months
  Capillarization will be determined using immunohistochemistry techniques
Change in skeletal muscle fiber typing | At baseline and at 6 months
  Fiber typing will be determined using immunohistochemistry techniques
Change in GLUT-4 protein expression | At baseline and at 6 months
  GLUT-4 protein expression will be assessed using immunoblotting techniques
Change reduced glutathione content in skeletal muscle cells | At baseline and at 6 months
  Reduced glutathione content will be determined spectrophotometrically
Change in glutathione peroxidase activity in skeletal muscle cells | At baseline and at 6 months
  Glutathione peroxidase activity will be determined spectrophotometrically
Change in glutathione reductase activity in skeletal muscle cells | At baseline and at 6 months
  Glutathione reductase activity will be determined spectrophotometrically
Change in superoxide dismutase activity in skeletal muscle cells | At baseline and at 6 months
  Superoxide dismutase activity will be determined spectrophotometrically
Change in fasting glucose levels | At baseline and at 6 months
  Fasting glucose levels will be measured on an automated clinical chemistry analyzer
Change in fasting insulin levels | At baseline and at 6 months
  Fasting insulin levels will be measured on an automated clinical chemistry analyzer
Change in glycosylated hemoglobin levels | At baseline and at 6 months
  Glycosylated hemoglobin levels will be measured on an automated clinical chemistry analyzer
Change in high-density lipoprotein (HDL) levels | At baseline and at 6 months
  HDL will be measured on an automated clinical chemistry analyzer
Change in low-density lipoprotein (LDL) levels | At baseline and at 6 months
  LDL will be measured on an automated clinical chemistry analyzer
Change in total cholesterol levels | At baseline and at 6 months
  Total cholesterol will be measured on an automated clinical chemistry analyzer
Change in triglyceride levels | At baseline and at 6 months
  Triglycerides will be measured on an automated clinical chemistry analyzer
Change in general blood count | At baseline and at 6 months
  General blood count will be measured on a hematology analyzer
Change in erythrocyte reduced glutathione (GSH) levels | At baseline and at 6 months
  Erythrocyte GSH levels will be determined spectrophotometrically
Change in erythrocyte oxidized glutathione (GSSG) levels | At baseline and at 6 months
  Erythrocyte GSSG levels will be determined spectrophotometrically
Change in myostatin expression | At baseline and at 6 months
  Myostatin expression will be assessed using immunoblotting techniques
Change cortisol concentration | At baseline and at 6 months
  Blood cortisol concentration will be assessed using immunoassays (ELISA)
Change in testosterone concentration | At baseline and at 6 months
  Blood testosterone concentration will be assessed using immunoassays (ELISA)
Change in growth hormone concentration | At baseline and at 6 months
  Blood growth hormone concentration will be assessed using immunoassays (ELISA)
Change in insulin-like growth factor-1 (IGF-1) concentration | At baseline and at 6 months
  Blood IGF-1 concentration will be assessed using immunoassays (ELISA)
Change in body mass | At baseline and at 6 months
  Body mass will be measured on a beam scale
Change in bone density | At baseline and at 6 months
  Bone density will be assessed using dual energy x-ray absorptiometry (DEXA)
Change in fat-free mass | At baseline and at 6 months
  Fat-free mass will be assessed using dual energy x-ray absorptiometry (DEXA)
Change in waist circumference | At baseline and at 6 months
  Waist circumference will be measured using a Gullick II tape
Change in hip circumference | At baseline and at 6 months
  Hip circumference will be measured using a Gullick II tape
Change in resting heart rate | At baseline and at 6 months
  Heart rate will be measured using a heart rate monitor
Change in resting metabolic rate (RMR) | At baseline and at 6 months
  RMR will be measured using indirect calorimetry
Change in systolic arterial pressure | At baseline and at 6 months
  Systolic blood pressure will be measured using a sphygmomanometer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Education and Sport Science Trikala, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided